CLINICAL TRIAL: NCT04777474
Title: Determination of Diagnostic Benefit of Enhanced Contact Endoscopy (ECE) in Pre-histological Diagnosis of Laryngeal and Hypopharyngeal Mucosal Lesions
Brief Title: Benefit of Enhanced Contact Endoscopy in Pre-histological Diagnosis of Laryngeal and Hypopharyngeal Mucosal Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23/RVO-FNOs/2020; 23/RVO-FNOs/2020 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2021-02-23; First posted 2021-03-02 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Laryngeal Disease; Laryngeal Lesions; Hypopharyngeal Lesions; Suspected Laryngeal Cancer; Suspected Hypopharyngeal Cancer; Proven Laryngeal Cancer; Proven Hypopharyngeal Cancer
Keywords: laryngeal cancer; hypopharyngeal cancer; laryngeal disease; enhanced contact endoscopy; narrow band imaging; IMAGE1S method
MeSH Terms: conditions — Laryngeal Diseases; Laryngeal Neoplasms; Hypopharyngeal Neoplasms | interventions — Narrow Band Imaging

STUDY DESIGN:
Intervention Model Description: The study subjects will be enrolled into one study group.
Masking Description: No masking is being used in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enhanced contact endoscopy (Experimental): The study subjects will undergo enhanced contact endoscopy
  Interventions: Diagnostic Test: Enhanced contact endoscopy; Diagnostic Test: Narrow band imaging; Diagnostic Test: IMAGE1S imaging

INTERVENTIONS:
Diagnostic Test: Enhanced contact endoscopy — The study subjects will undergo enhanced contact endoscopy - studied imaging technique
Diagnostic Test: Narrow band imaging — The study subjects will undergo narrow band imaging - comparator procedure
Diagnostic Test: IMAGE1S imaging — The study subjects will undergo IMAGE1S imaging - comparator procedure

SUMMARY:
The focus of the study is to verify the role of enhanced contact endoscopy in early identification of high-risk vascular patterns of precancerous and malignant mucosal changes in ear-nose-throat (ENT) patients, in comparison with other standard imaging techniques.

DETAILED DESCRIPTION:
Endoscopy methods are inseparable part in diagnostics of patients with head and neck cancer. Nowadays ENT surgeons are offered a wide variety of endoscopy methods. The methods that caused revolution in early diagnostics of head and neck cancer were advanced imagining endoscopy methods such as NBI or IMAGE1S.

The new only recently introduced method is enhanced contact endoscopy, which uses a combination of advanced imagining, such as NBI or IMAGE1S, with rigid microlaryngoscope. It is believed that this technology has the potential to visualise vascular patterns of precancerous and malignant mucosal changes even better than narrow-band imaging (NBI) and IMAGE1S. This improvement in diagnostics helps with early identification of high-risk lesions and moves us closer to the concept of pre-histological diagnostics, which helps to accelerate making final diagnosis, which leads to prompt treatment.

Study protocol:

* anamnestic questionnaire (age, sex, weight, height, smoking, alcohol, reflux disease)
* Reflux Symptom Index (RSI) questionnaire
* endoscopy in white light in local anaesthesia with evaluation:
* character of the lesion (benign, Reinke edema, cyst, polyp, chronic laryngitis/pharyngitis, leukoplakia, erythroplakia, malignity)
* bleeding or ulceration on the surface of the lesion
* endoscopy with NBI endoscope in local anesthesia with evaluation:
* mucosa vascularization according to the ELS classification
* size of the lesion in compare to endoscopy in white light in local anesthesia
* occurrence of new lesions in compare to endoscopy in white light in local anesthesia
* endoscopy in white light in general anesthesia during microlaryngoscopy
* character of the lesion (benign, Reinkes edema, cyst, polyp, chronic laryngitis/pharyngitis, leukoplakia, erythroplakia, malignity)
* bleeding or ulceration on the surface of the lesion
* size of the lesion in compare to endoscopy in white light in local anesthesia
* occurence of new lesions when compared with endoscopy in white light in local anesthesia
* endoscopy in NBI or IMAGE1S in general anesthesia during microlaryngoscopy
* mucosa vascularization according to the ELS classification
* size of the lesion in compare to endoscopy in white light in local anesthesia
* occurence of new lesions in compare to endoscopy in white light in local anesthesia
* enhanced contact endoscopy (ECE) in NBI or IMAGE1S in general anesthesia during microlaryngoscopy
* mucosa vascularization according to the ELS and Puxxedu classification
* size of the lesion in compare to endoscopy in white light and NBI/ IMAGE1S in general anesthesia
* occurence of new lesions in compare to endoscopy in white light and NBI/

IMAGE1S in general anesthesia

* histology examination with determination of final diagnosis
* benign lesion
* mild dysplasia
* severe dysplasia
* carcinoma in situ
* invasive cancer

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* patients scheduled for direct hypopharyngoscopy and laryngoscopy in general anaesthesia
* benign laryngeal and hypoharyngeal disease/laryngeal and hypopharyngeal lesions of uncertain biologic behaviour (leukoplakia, erythroplakia, keratosis)
* patients with suspicious macroscopical lesion found during ENT examination/patients with histologically confirmed metastasis of carcinoma in neck lymph node with unknown primary origin of the tumour
* patients with recurrence of malign tumour in hypopharynx or larynx
* patients after radiotherapy indicated for follow up examination under general anaesthesia
* patients with persistent non-specific problems (hoarseness, swallowing problems etc.) indicated to direct laryngohypopharyngoscopy due to diagnostic purposes

Exclusion Criteria:

* age - younger than 17 years
* refusal to join the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of enhanced contact endoscopy | Procedure (During the examination under general anaesthesia)
  The accuracy of enhanced contact endoscopy will be observed (size of lesions in mm when compared with the other standard techniques)
Sensitivity of enhanced contact endoscopy | Procedure (During the examination under general anaesthesia)
  The sensitivity of enhanced contact endoscopy in making pre-histological diagnosis using final histopathology result. will be observed.
Specificity of enhanced contact endoscopy | Procedure (During the examination under general anaesthesia)
  The specificity of enhanced contact endoscopy in making pre-histological diagnosis using final histopathology result. will be observed.
Positive predictive value of enhanced contact endoscopy | Procedure (During the examination under general anaesthesia)
  The positive predictive value of enhanced contact endoscopy in making pre-histological diagnosis using final histopathology result. will be observed.
Negative predictive value of enhanced contact endoscopy | Procedure (During the examination under general anaesthesia)
  The negative predictive value of enhanced contact endoscopy in making pre-histological diagnosis using final histopathology result. will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kántor, MD, Principal Investigator — University Hospital Ostrava
Locations (2):
- Czechia (2):
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region
  - University Hospital Hradec Králové, Hradec Králové

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Background] Puxeddu R, Sionis S, Gerosa C, Carta F. Enhanced contact endoscopy for the detection of neoangiogenesis in tumors of the larynx and hypopharynx. Laryngoscope. 2015 Jul;125(7):1600-6. doi: 10.1002/lary.25124. Epub 2015 Jan 13. PMID 25582112
- [Background] Mehlum CS, Dossing H, Davaris N, Giers A, Grontved AM, Kjaergaard T, Moller S, Godballe C, Arens C. Interrater variation of vascular classifications used in enhanced laryngeal contact endoscopy. Eur Arch Otorhinolaryngol. 2020 Sep;277(9):2485-2492. doi: 10.1007/s00405-020-06000-z. Epub 2020 Apr 30. PMID 32350646